CLINICAL TRIAL: NCT02424227
Title: Circulating Donor-Derived Cell-free DNA in Blood for Diagnosing Acute Rejection in Kidney Transplant Recipients
Brief Title: Non Invasive Blood Test To Diagnose Acute Rejection After Kidney Transplantation
Acronym: DART
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: CareDx (Industry)
Responsible Party: Sponsor
Other Study IDs: SN-C-00006
Record Dates: First submitted 2015-04-20; First posted 2015-04-22 (Estimated); Last update posted 2018-12-17 (Actual); Status verified 2018-12

CONDITIONS: Kidney Transplant Recipients

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — cfDNA samples collected in Cell-Free DNA BCT and mRNA collected in PAX gene tubes will be retained
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Kidney Transplant Recipients: Adult living and deceased donor kidney transplant recipients will be eligible to participate in this study.

SUMMARY:
This is a prospective, multicenter, observational study of kidney transplant subjects where blood specimens, intended for dd-cfDNA and other future research purposes, will be drawn after transplant

DETAILED DESCRIPTION:
This is a prospective, multicenter, observational study of kidney transplant subjects where blood specimens, intended for dd-cfDNA and other future research purposes, will be drawn after transplant periodically and also after the treatment of acute rejection up to 8 weeks post treatment. The blood samples and all relevant clinical data will be provided to CareDx scientists for laboratory assay of dd-cfDNA levels and correlation of dd-cfDNA levels with the clinical features of the subjects.

The primary objective of the study is to correlate circulating dd-cfDNA to clinical and sub-clinical acute rejection in renal allograft recipients. The secondary objective of the study is to correlate circulating dd-cfDNA to renal function, both serum creatinine and estimated glomerular filtration rate [eGFR]).

ELIGIBILITY:
Inclusion Criteria

1. Adult recipients (Age > 18 years )
2. Both genders and all racial and ethnic groups
3. Kidney transplant alone
4. Both living and deceased donor transplants
5. Primary and re-transplants. A total of 30 re-transplant recipients across all study sites will be eligible for enrollment. CareDx will notify all centers when this subset of enrollment has been met. Thereafter, all enrolled patients should be primary transplant recipients.
6. Ability to come for follow-up and undergo biopsy (Performed in accordance to SOC)
7. Ability to give written informed consent prior to study enrollment

Patients can be enrolled at any time; before or after transplantation and/or at time of outpatient or inpatient visits for workup of medical problems; e.g. at the time of a renal biopsy (regardless of elapsed time since post transplant) as specified in this study protocol.

Exclusion Criteria

1. Pediatric recipients (Age < 18 years)
2. Pregnant women
3. Patients undergoing multi-organ transplants (e.g. kidney with pancreas or liver)
4. Patients receiving donor organ from an identical twin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult de novo living and deceased donor kidney transplant recipients will be eligible to participate in this study.
Sampling Method: Non-Probability Sample
Enrollment: 401 (Actual)
Dates: Start 2015-04; Primary Completion 2018-08-30 (Actual); Study Completion 2019-01-31 (Estimated)

PRIMARY OUTCOMES:
Clinical T cell as well as antibody mediated acute rejection | Occurring within 12 months post transplant
Sub-clinical T cell as well as antibody mediated acute rejection | Occurring within 12 months post transplant
Composite of clinical and sub-clinical T cell as well as antibody mediated acute rejection | Occurring within 12 months post transplant

SECONDARY OUTCOMES:
eGFR (estimated Glomerular Filtration Rate [mL/min]): will be derived from serum creatinine level, corrected for variables, using the CKD-RPI (Chronic Kidney Disease Epidemiology Collaboration) equation | 24 months
Renal allograft injury from BKV nephritis, CNI toxicity, acute pyeloenephrtiis and recurrent disease confirmed by renal histology | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: James Yee, MD, Study Director — CareDx
Locations (14):
- United States (14):
  - University of Alabama, Birmingham, Birmingham, Alabama
  - University of California Los Angeles, Los Angeles, California
  - Cedars-Sinai Medical Center, Los Angeles, California
  - Indiana University, Indianapolis, Indiana
  - University of Maryland, Baltimore, Maryland
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University, St Louis, Missouri
  - Columbia University, New York, New York
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of Pennsylvannia, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - Baylor Research Institute, Fort Worth, Texas
  - Baylor Scott and White, Temple, Texas

REFERENCES:
- [Background] Haas M, Sis B, Racusen LC, Solez K, Glotz D, Colvin RB, Castro MC, David DS, David-Neto E, Bagnasco SM, Cendales LC, Cornell LD, Demetris AJ, Drachenberg CB, Farver CF, Farris AB 3rd, Gibson IW, Kraus E, Liapis H, Loupy A, Nickeleit V, Randhawa P, Rodriguez ER, Rush D, Smith RN, Tan CD, Wallace WD, Mengel M; Banff meeting report writing committee. Banff 2013 meeting report: inclusion of c4d-negative antibody-mediated rejection and antibody-associated arterial lesions. Am J Transplant. 2014 Feb;14(2):272-83. doi: 10.1111/ajt.12590. PMID 24472190
- [Background] Lo YM. Transplantation monitoring by plasma DNA sequencing. Clin Chem. 2011 Jul;57(7):941-2. doi: 10.1373/clinchem.2011.166686. No abstract available. PMID 21566070
- [Background] Snyder TM, Khush KK, Valantine HA, Quake SR. Universal noninvasive detection of solid organ transplant rejection. Proc Natl Acad Sci U S A. 2011 Apr 12;108(15):6229-34. doi: 10.1073/pnas.1013924108. Epub 2011 Mar 28. PMID 21444804
- [Background] Code of Federal Regulations, Title 42 - Public Health, Part 493 - Laboratory Requirements, Subpart A - General Provisions, Sections 1, 2 & 3
- [Background] Hidestrand M, Tomita-Mitchell A, Hidestrand PM, Oliphant A, Goetsch M, Stamm K, Liang HL, Castleberry C, Benson DW, Stendahl G, Simpson PM, Berger S, Tweddell JS, Zangwill S, Mitchell ME. Highly sensitive noninvasive cardiac transplant rejection monitoring using targeted quantification of donor-specific cell-free deoxyribonucleic acid. J Am Coll Cardiol. 2014 Apr 1;63(12):1224-1226. doi: 10.1016/j.jacc.2013.09.029. Epub 2013 Oct 16. No abstract available. PMID 24140666
- [Background] Sigdel TK, Vitalone MJ, Tran TQ, Dai H, Hsieh SC, Salvatierra O, Sarwal MM. A rapid noninvasive assay for the detection of renal transplant injury. Transplantation. 2013 Jul 15;96(1):97-101. doi: 10.1097/TP.0b013e318295ee5a. PMID 23756769
- [Background] De Vlaminck I, Valantine HA, Snyder TM, Strehl C, Cohen G, Luikart H, Neff NF, Okamoto J, Bernstein D, Weisshaar D, Quake SR, Khush KK. Circulating cell-free DNA enables noninvasive diagnosis of heart transplant rejection. Sci Transl Med. 2014 Jun 18;6(241):241ra77. doi: 10.1126/scitranslmed.3007803. PMID 24944192
- [Derived] Sawinski DL, Mehta S, Alhamad T, Bromberg JS, Fischbach B, Aeschbacher T, Ghosh S, Shekhtman G, Dholakia S, Brennan DC, Poggio E, Bloom RD, Jordan SC. Association between dd-cfDNA levels, de novo donor specific antibodies, and eGFR decline: An analysis of the DART cohort. Clin Transplant. 2021 Sep;35(9):e14402. doi: 10.1111/ctr.14402. Epub 2021 Jul 14. PMID 34184326
- [Derived] Bromberg JS, Brennan DC, Poggio E, Bunnapradist S, Langone A, Sood P, Matas AJ, Mannon RB, Mehta S, Sharfuddin A, Fischbach B, Narayanan M, Jordan SC, Cohen DJ, Zaky ZS, Hiller D, Woodward RN, Grskovic M, Sninsky JJ, Yee JP, Bloom RD. Biological Variation of Donor-Derived Cell-Free DNA in Renal Transplant Recipients: Clinical Implications. J Appl Lab Med. 2017 Nov 1;2(3):309-321. doi: 10.1373/jalm.2016.022731. PMID 33636851